CLINICAL TRIAL: NCT03818386
Title: Radiotherapy of Multiple Brain Metastases Using AGuIX® Gadolinium-chelated Polysiloxane Based Nanoparticles: a Prospective Randomized Phase II Clinical Trial.
Brief Title: Radiotherapy of Multiple Brain Metastases Using AGuIX®
Acronym: NANORAD2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: NH TherAguix SAS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 38RC18.085
Record Dates: First submitted 2018-12-11; First posted 2019-01-28 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2023-08

CONDITIONS: Brain Metastases, Adult; Radiotherapy
Keywords: gadolinium nanoparticles; AGuIX
MeSH Terms: conditions — Brain Neoplasms | interventions — AGuIX

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Open Blinded Endpoint phase II clinical trial.
Who Masked: Outcomes Assessor
Masking Description: The main endpoint will be evaluated by a blinded endpoint committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AGuIX® + Whole Brain Radiation Therapy (Experimental): Intervention: Drug: AGuIX® + WBRT
  Other Names:
  Gadolinium-chelated polysiloxane based nanoparticles
  3 intravenous injections at 100mg/kg
  * D0: AGuIX® injection followed by MRI (within 7 days before commencement of WBRT)
  * Fr1: AGuIX® injection before the first radiation session
  * Fr6: AGuIX® injection before the sixth radiation session
    30 Gy in 10 fractions of 3 Gy over 2-3 weeks
  Interventions: Drug: AGuIX®; Radiation: Whole Brain Radiation Therapy
- Whole Brain Radiation Therapy (Active Comparator): Intervention: Radiation: Whole Brain Radiation Therapy ( WBRT) 30 Gy in 10 fractions of 3 Gy over 2-3 weeks
  Interventions: Radiation: Whole Brain Radiation Therapy

INTERVENTIONS:
Drug: AGuIX® — 3 intravenous injection at 100mg/kg
  * D0: AGuIX® injection followed by MRI (within 7 days before commencement of WBRT)
  * Fr1: AGuIX® injection before the first radiation session
  * Fr6: AGuIX® injection before the sixth radiation session
  Other Names: Gadolinium-chelated polysiloxane based nanoparticles
  Arms: AGuIX® + Whole Brain Radiation Therapy
Radiation: Whole Brain Radiation Therapy — 30 Gy in 10 fractions of 3 Gy over 2-3 weeks
  Other Names: WBRT

SUMMARY:
This is a Prospective Randomized Open Blinded Endpoint phase II clinical trial. The study will be adaptive: an interim analysis is planned after enrolment of 20 patients in each arm of treatment (WBRT and AGuIX® + WBRT), to select and continue the study with group(s) that present the best response rate to the experimental treatment (AGuIX® + WBRT).

The main endpoint will be evaluated by a blinded endpoint committee.

DETAILED DESCRIPTION:
The occurrence of brain metastases is a common event in the history of cancer and negatively affects the life expectancy of patients. Their incidence varies between 15 and 50% according to the histologic types. Surgery, stereotactic radiosurgery, radiotherapy and chemotherapy are the main treatments currently proposed.

For patients with multiple brain metastases, whole brain radiation therapy (WBRT) remains the standard of care. However, the median overall survival is less than 6 months and new approaches need to be developed to improve treatment of these patients.

In this context, the weak control of the disease comes from three main factors: the multiplicity of the brain lesions, the radioresistance of certain histologies and the poor distribution of cytotoxic agents in brain metastases.

The use of radiosensitizing agents is here of great interest. The radiosensitizing agent chosen in this study is AGuIX®. It is a Gadolinium-chelated polysiloxane based nanoparticle developed by NH TherAguix company for its theranostic properties (radiosensitization and diagnosis by multimodal imaging). Preclinical studies have demonstrated the radiosensitizing effect of AGuIX® in vivo in 8 tumor models xenografted in rodents, and particularly in brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with brain metastases, from a histologically confirmed solid tumor, eligible for WBRT
* At least 18 years old
* Signed informed consent after informing the patient
* ECOG (Eastern Cooperative Oncology Group) performance status 0-2
* Extracranial disease:

  * Complete or partial response or stability under systemic treatment
  * No extracranial disease
  * Or first line of treatment
* Life expectancy greater than 6 weeks
* Effective contraceptive method for all patient of childbearing potential
* Affiliated to a social security regimen

Exclusion Criteria:

* Leptomeningeal metastasis
* Evidence of metastasis with recent large hemorrhage
* Progressive and threatening extracranial disease under systemic treatment
* Previous cranial irradiation (except stereotactic irradiation)
* Known contra-indication, sensitivity or allergy to gadolinium
* Known contra-indication for Magnetic Resonance Imaging
* Renal insufficiency (glomerular filtration rate ≤ 50 mL/min/1.73m²)
* Pregnancy or breastfeeding
* Subject under administrative or judicial control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-03-26 (Actual); Primary Completion 2024-06-26 (Estimated); Study Completion 2025-03-26 (Estimated)

PRIMARY OUTCOMES:
Best objective intracranial response rate - intent-to-treat | at 6 weeks
  Evaluation of brain metastases response, according to RECIST v1.1 criteria (or modified RECIST) by MRI, with MRI centralized reading
Best objective intracranial response rate - intent-to-treat | at 3 months
  Evaluation of brain metastases response, according to RECIST v1.1 criteria (or modified RECIST) by MRI, with MRI centralized reading

SECONDARY OUTCOMES:
Evaluation of the quality of life | at D0, 6 weeks, 3, 6, 9, 12 months
  Quality of life test score EORTC QLQ C30
Evaluation of the quality of life | at day 0, 6 weeks, 3, 6, 9, 12 months
  Quality of life test score EORTC QLQ BN20
Neurocognitive evaluation | at Day 0, 6 weeks, 3, 6, 9, 12 months
  Neurocognitive test (MoCA)
Best objective intracranial response rate - per-protocol | at 6 weeks and 3 months
  Evaluation of brain metastases response on per-protocol population, according to RECIST v1.1 criteria (or modified RECIST), by MRI with centralized reading
Evaluation of the intracranial response rate | for 12 months
  Evaluation of brain metastases response, according to RANO, to RECIST v1.1 criteria, and as the evolution of the sum of longest diameters (for all metastases with a sum of diameters > 1cm), by MRI, at 6 weeks and 3, 6, 9 and 12 months
Evaluation of individual metastasis response | at 6 weeks and 3, 6, 9 and 12 months
  Evaluation of individual brain metastasis response, for all metastases with the sum of diameters > 1cm, by MRI rate
Intracranial progression-free survival | at 12 months
  Evaluation of the time between the start of the treatment and the occurence of intracranial progression or neuriologic death
Intracranial progression-free survival, brain survival | at 12 months
  Death related to brain metastases progression
Overall survival | at 12 months
  Death
Change in steroid dependence | at 6 weeks and 3, 6, 9 and 12 months
  Reporting of daily steroid dose
Incidence of adverse events | at 6 weeks and 3, 6, 9 and 12 months
  Reporting of adverse events by type, frequency and severity for both treatments (WBRT and AGuIX® + WBRT)
MRI study of the distribution of the product in brain metastases | Day 0
  MRI evaluation of contrast enhancement at D0 after AGuIX® injection

CONTACTS AND LOCATIONS:
Overall Officials: Camille VERRY, MD, Principal Investigator — University Hospital, Grenoble
Locations (14):
- France (14):
  - Institut Régional du Cancer, Montpellier, Occitanie
  - Institut Claudius Regaud Institut Universitaire du Cancer Toulouse Oncopole Radiothérapie, Toulouse, Occitanie
  - Centre Leon Berard Lyon, Lyon, Rhones Alpes
  - Centre Hospitalier Annecy Genevois, Annecy, Rhones-Alpes
  - Centre Hospitalier Universitaire Grenoble-Alpes, Grenoble, Rhones-Alpes
  - CRLCC - Institut Bergonié, Bordeaux
  - Crlcc Francois Baclesse, Caen
  - Centre Georges François Leclerc, Dijon
  - Hospices Civils de Lyon-Hôpital Lyon Sud, Lyon
  - Hôpital Européen Georges Pompidou, Paris
  - La Pitié Salpêtrière - Charles Foix, Paris
  - Institut Curie Saint Cloud, Saint-Cloud
  - Crlcc Paul Strauss, Strasbourg
  - Institut de Cancérologie de Lorraine ALEXIS VAUTRIN, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le Duc G, Miladi I, Alric C, Mowat P, Brauer-Krisch E, Bouchet A, Khalil E, Billotey C, Janier M, Lux F, Epicier T, Perriat P, Roux S, Tillement O. Toward an image-guided microbeam radiation therapy using gadolinium-based nanoparticles. ACS Nano. 2011 Dec 27;5(12):9566-74. doi: 10.1021/nn202797h. Epub 2011 Nov 9. PMID 22040385
- [Background] Lux F, Tran VL, Thomas E, Dufort S, Rossetti F, Martini M, Truillet C, Doussineau T, Bort G, Denat F, Boschetti F, Angelovski G, Detappe A, Cremillieux Y, Mignet N, Doan BT, Larrat B, Meriaux S, Barbier E, Roux S, Fries P, Muller A, Abadjian MC, Anderson C, Canet-Soulas E, Bouziotis P, Barberi-Heyob M, Frochot C, Verry C, Balosso J, Evans M, Sidi-Boumedine J, Janier M, Butterworth K, McMahon S, Prise K, Aloy MT, Ardail D, Rodriguez-Lafrasse C, Porcel E, Lacombe S, Berbeco R, Allouch A, Perfettini JL, Chargari C, Deutsch E, Le Duc G, Tillement O. AGuIX(R) from bench to bedside-Transfer of an ultrasmall theranostic gadolinium-based nanoparticle to clinical medicine. Br J Radiol. 2019 Jan;92(1093):20180365. doi: 10.1259/bjr.20180365. Epub 2018 Sep 18. PMID 30226413
- [Background] Verry C, Dufort S, Barbier EL, Montigon O, Peoc'h M, Chartier P, Lux F, Balosso J, Tillement O, Sancey L, Le Duc G. MRI-guided clinical 6-MV radiosensitization of glioma using a unique gadolinium-based nanoparticles injection. Nanomedicine (Lond). 2016 Sep;11(18):2405-17. doi: 10.2217/nnm-2016-0203. Epub 2016 Aug 16. PMID 27529506